CLINICAL TRIAL: NCT07167251
Title: Management of Immune Checkpoint Inhibition-related Hepatitis Using Low-dose Corticosteroids - A Prospective Registry-based, Cohort Study
Brief Title: Management of Immune Checkpoint Inhibition-related Hepatitis Using Low-dose Corticosteroids
Acronym: MIRA-HEP
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Royal Marsden NHS Foundation Trust (Other); Odense University Hospital (Other); UMC Utrecht (Other)
Responsible Party: Principal Investigator, Andreas Schmitt, Deputy Physician, University Hospital, Basel, Switzerland
Other Study IDs: 2025-00696
Record Dates: First submitted 2025-08-25; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Immune Related Adverse Events; Immune-Mediated Hepatitis; Cancer
Keywords: Immune-related adverse events; Immune checkpoint inhibitor; Immune-related hepatitis; immune-mediated hepatitis
MeSH Terms: conditions — Neoplasms | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Immune-related hepatitis grade 2: Grade 2 hepatitis is defined as an elevation of Aspartate transaminase (AST) and/or Alanine aminotransferase (ALT) levels to 3-5 times the upper limit of normal, in accordance with the guidelines of the European Society for Medical Oncology.
  Interventions: Drug: Low-dose corticosteroids for immune-related hepatitis grade 2
- Immune-related hepatitis grade 3: Grade 3 hepatitis is defined as an elevation of Aspartate transaminase and/or Alanine aminotransferase levels to 5-20 times the upper limit of normal, in accordance with the guidelines of the European Society for Medical Oncology.
  Interventions: Drug: Low-dose corticosteroids for immune-related hepatitis grade 3

INTERVENTIONS:
Drug: Low-dose corticosteroids for immune-related hepatitis grade 3 — Prednisolone 0.5-1 mg/kg orally for grade 3 IR-hepatitis; adjusted based on liver function; treatment per local standard of care.
  Groups: Immune-related hepatitis grade 3
Drug: Low-dose corticosteroids for immune-related hepatitis grade 2 — Hold immunotherapy and reassess liver function at the treating physician's discretion. If liver function tests persistently worsen or continue to rise, consider administering prednisolone at 0.5 mg/kg body weight
  Groups: Immune-related hepatitis grade 2

SUMMARY:
This study evaluates the effectiveness of low-dose corticosteroids in managing grade 2-3 immune-related hepatitis in cancer patients treated with immune checkpoint inhibitors. It aims to determine whether of 0.5-1miligram per kilogram bodyweight prednisolone is sufficient to manage immune-related hepatitis without the need for dose escalation or additional immunosuppressive therapy.

DETAILED DESCRIPTION:
Immune checkpoint inhibitors (ICIs) have revolutionized cancer therapy but are associated with immune-related adverse events (irAEs), including immune-related hepatitis, a potentially serious complication that affects up to 30% of patients undergoing ICI combination therapy. Current management guidelines recommend corticosteroids as the first-line treatment for moderate to severe irAEs. However, high doses of corticosteroids are associated with increased risks of infections, metabolic and psychiatric side effects, and potentially impaired anti-tumor efficacy. Retrospective data suggest that lower doses may be equally effective while reducing toxicity and preserving treatment efficacy.

This prospective, registry-based cohort study aims to evaluate the clinical performance and outcomes of low-dose corticosteroid treatment for managing grade 2 or 3 IR-hepatitis. The hypothesis is that a corticosteroid "test dose" approach (0.5-1 mg/kg prednisolone) followed by early evaluation of clinical response can identify patients who benefit from reduced immunosuppression, thus minimizing side effects without compromising the effectiveness of ICI therapy.

Patients will be recruited from participating oncology centers where standardized management of IR-hepatitis has been implemented. Eligible participants are adult cancer patients who develop grade 2 or 3 IR-hepatitis during ICI therapy, excluding those with prior high-dose corticosteroid use, concurrent neurological or cardiac irAEs requiring high-dose corticosteroids, or underlying chronic liver diseases.

The primary endpoint is resolution of IR-hepatitis (defined as return to baseline or grade 1 liver function tests) within 8 weeks without corticosteroid dose escalation, additional immunosuppressive therapy, and with tapering to ≤10 mg/day prednisolone. Secondary endpoints include the proportion of patients requiring dose escalation, time to hepatitis resolution, cumulative corticosteroid exposure, relapse rates, occurrence of additional irAEs, progression-free survival (PFS), overall survival (OS), and identification of predictors of steroid-refractory hepatitis.

Patients will be followed for six months after the onset of IR-hepatitis. Follow-up assessments will align with standard clinical care, with no additional study-specific visits. Liver function tests, immunotherapy status, corticosteroid and immunosuppressive use, and occurrence of new irAEs will be recorded. A liver biopsy is recommended in refractory or ambiguous cases. Data will be collected via the REDCap system, ensuring standardized electronic data capture.

The study is powered to detect a successful resolution rate of at least 80% in patients with grade 3 IR-hepatitis treated with low-dose corticosteroids, assuming a null hypothesis threshold of 65%. Descriptive and exploratory statistical methods will be used to analyze the data, including Kaplan-Meier estimates for time-to-event outcomes and logistic regression for exploratory subgroup analyses.

This study addresses a critical gap in prospective evidence on the management of IR-hepatitis. By evaluating the efficacy and safety of a pragmatic, low-cost, low-toxicity intervention, it may inform future guidelines and serve as a foundation for a randomized non-inferiority trial. The study's design allows for real-world applicability while ensuring scientific rigor through harmonized protocols and data collection.

ELIGIBILITY:
Inclusion Criteria:

1. Cancer patients aged 18 years or older
2. Treatment with a programmed cell death protein 1 (PD-1) or programmed cell death ligand 1 (PD-L1) antibody, or a cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) antibody, or a combination of a PD-1 and CTLA-4 antibody, or a PD-1 and lymphocyte-activation gene 3 (LAG-3) antibody
3. Occurrence of immune-related hepatitis grade 2 to 3 (as per judgment of the investigator)
4. Ability of the patient to comply with the study procedures (management of immune-related hepatitis)

Exclusion Criteria:

1. Previous Immune-related hepatitis that required systemic therapy
2. Treatment for Immune-related hepatitis has already been initiated with high-dose corticosteroids (>0.5 mg/kg body weight)
3. Immune-related hepatitis with bilirubin > 1.5 ULN or clinical suspicion of cholangitis or elevated INR (beyond baseline)
4. Immune-related hepatitis with grade 4 at first presentation
5. Prior irAE treated with systemic immunosuppression
6. Simultaneous immune-related neurological toxicity or immune-related myocarditis (since these usually have to be treated with high doses of corticosteroids)

   a. Patients with other immune-related adverse events may be included according to the investigator's judgment
7. Known liver disease (e.g., autoimmune hepatitis, active hepatitis B, C or E, hemochromatosis, liver cirrhosis Child-Pugh Score B or C, primary biliary cholangitis, primary biliary cirrhosis, Morbus Wilson)

   a. Patients with liver metastasis are eligible
8. Patients receiving cancer treatment other than immune checkpoint inhibitors in parallel (e.g., tyrosine kinase inhibitors or chemotherapy).

   a. Patients who have received other cancer treatments in previous cycles are eligible, provided the treating physician does not assume any toxicity from the other medication.
9. Condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications within 14 days prior to occurrence of IR hepatitis. Stable corticosteroid doses of < 10mg prednisone equivalent are allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target patient population of this study are patients treated with immune checkpoint inhibitors (either as monotherapy with an anti-programmed cell death protein 1 (PD-1) or programmed cell death ligand 1 (PD-L1) antibody, or with an anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) antibody, or as combination therapy with an PD-1 and CTLA-4 antibody, or an PD-1 and lymphocyte-activation gene 3 (LAG3) antibody) who develop grade 2 or 3 Immune-related hepatitis independently of the treated cancer entity.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with resolution of their IR hepatitis CTCAE grade 3 within 8 weeks of onset | 8 weeks of onset
  Resoultion is defined as back to baseline or grade 1 without escalation of the corticosteroid dose, without additional immunosuppression and with discontinuation of corticosteroids or reduction to a maximum of 10 mg of Prednisolone

SECONDARY OUTCOMES:
Proportion of patients with resolution of their IR hepatitis CTCAE grade 2 or 3 within 8 weeks of onset | 8 weeks
  Resoultion is defined as back to baseline or grade 1 without escalation of the corticosteroid dose, without additional immunosuppression and with discontinuation of corticosteroids or reduction to a maximum of 10 mg of Prednisolone
Proportion of patients requiring dose escalation of corticosteroids | Outcome assessed at each visit until end of follow-up (6 months).
Time to resolution of IR hepatitis | Outcome assessed at each visit until end of follow-up (6 months).
Peak dose of corticosteroids | Outcome assessed at each visit until end of follow-up (6 months).
  Maximum dose of corticosteroids used for the treatment of IR hepatitis
Cumulative dose of corticosteroids | Outcome assessed at each visit until end of follow-up (6 months).
  Cumulative dose of corticosteroids used for the treatment of IR hepatitis
Proportion of patients with relapse of their IR hepatitis to grade 2 or higher | Outcome assessed at each visit until end of follow-up (6 months).
Proportion of patients with incidence of irAE other than IR hepatitis | Outcome assessed at each visit until end of follow-up (6 months).
Progression-free survival | Up to 6 months
  Time from first registration until the first documented disease progression, or death from any cause, whichever occurs first. Participants without an event will be censored at the date of last disease assessment.
Overall survival | Up to 6 months
  Time from first registration until death from any cause. Participants who are alive at last follow-up will be censored at the date of last contact.
Association of patient, disease and treatment characteristics and occurrence of corticosteroid refractory IR hepatitis | Patient, disease and treatment characteristics at baseline

OTHER OUTCOMES:
Recruitment rate | At recruitment completion (last patient enrolled, up to 18 months)
  Number of registered patients per months
Retention rate | At study completion (final follow-up, 6 months after inclusion of the last patient])
  The number and proportion of patients with a complete follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Andreas M Schmitt, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (2):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland
- Royal Marsden Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data (IPD) will be available on request from qualified researchers after publication.
Supporting Information: Study Protocol